CLINICAL TRIAL: NCT00281346
Title: Non-invasive Evaluation of Coronary Pathology by Transthoracic Doppler Echocardiography. A Comparative Study to Coronary Angiography.
Brief Title: Non-invasive Diagnosis of Coronary Artery Stenoses by Doppler Echocardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29 FU-71-05
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Stable Angina Pectoris; Unstable Angina Pectoris; Acute Myocardial Infarction
Keywords: Doppler echocardiography; coronary stenosis; Coronary angiography
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- transthoracic Doppler echocardiography (Experimental)
  Interventions: Procedure: Doppler echocardiography

INTERVENTIONS:
Procedure: Doppler echocardiography — Echocardiography

SUMMARY:
Non-invasive evaluation of patients with stable angina and unstable coronary syndromes with transthoracic Doppler echocardiography to evaluate presence of significant coronary stenoses. Blinded evaluation and comparison with coronary angiography: presence and location of stenoses, and head to head comparison of clinical value and patient classification.

DETAILED DESCRIPTION:
Transthoracic Doppler echocardiographic evaluation with extensive evaluation of coronary stenoses in all 3 main branches using colour flow, pulsed Doppler and Coronary flow velocity reserve (CFVR)after pharmacologic stress with adenosin in the area of LAD and RDP. Blinded evaluation of Doppler results and coronary angiography regarding the other examination modality. Coronary angiography diagnostic "gold standard". Only stable and unstable patients otherwise scheduled for angiography on clinical reasons will be examined and included in the study.

Added January 2007 after ethics committee approval: comparison of CFVR with invasive fractional flow reserve (FFR) in selected subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* unstable angina or acute myocardial infarction, or stable angina pectoris and
* scheduled for coronary angiography on accepted clinical reasons

Exclusion Criteria:

* past coronary artery grafting

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield: Accuracy, positive and negative predictive value. | Inhospital
pr patient evaluation | Inhospital

SECONDARY OUTCOMES:
pr stenosis evaluation | Inhospital

CONTACTS AND LOCATIONS:
Overall Officials: Torstein L Hole, MD, PhD, Study Chair — Norwegian University of Science and Technology; Johnny Å Vegsundvåg, MD, Principal Investigator; Rune Wiseth, MD, PhD, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Ålesund Hospital HF, Ålesund, Norway

REFERENCES:
- [Result] Holte E, Vegsundvag J, Hegbom K, Hole T, Wiseth R. Transthoracic Doppler for detection of stenoses in the three main coronary arteries by use of stenotic to prestenotic velocity ratio and aliased coronary flow. Eur Heart J Cardiovasc Imaging. 2015 Dec;16(12):1323-30. doi: 10.1093/ehjci/jev158. Epub 2015 Jun 25. PMID 26113119
- [Derived] Vegsundvag J, Holte E, Wiseth R, Hegbom K, Hole T. Coronary artery occlusions diagnosed by transthoracic Doppler. Cardiovasc Ultrasound. 2014 Mar 15;12:12. doi: 10.1186/1476-7120-12-12. PMID 24628779
- [Derived] Vegsundvag J, Holte E, Wiseth R, Hegbom K, Hole T. Coronary flow velocity reserve in the three main coronary arteries assessed with transthoracic Doppler: a comparative study with quantitative coronary angiography. J Am Soc Echocardiogr. 2011 Jul;24(7):758-67. doi: 10.1016/j.echo.2011.03.010. Epub 2011 Apr 23. PMID 21524564
- [Derived] Vegsundvag J, Holte E, Wiseth R, Hegbom K, Hole T. Transthoracic echocardiography for imaging of the different coronary artery segments: a feasibility study. Cardiovasc Ultrasound. 2009 Dec 22;7:58. doi: 10.1186/1476-7120-7-58. PMID 20028530